CLINICAL TRIAL: NCT04019496
Title: Neurophysiological Characterization of Treatment Response Following the Initiation of Prophylactic Therapy in Episodic Migraine
Brief Title: Neurophysiology of Prophylactic Treatment in Migraine
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB168/18
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Migraine
Keywords: blink reflex; electroencephalography; functional magnetic resonance imaging; evoked potentials
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic Migraine
  Interventions: Drug: antibodies against calcitonin-gene related peptide or its receptor
- Healthy controls: equal to or less than 1 headache day/month

INTERVENTIONS:
Drug: antibodies against calcitonin-gene related peptide or its receptor — the study is observational and does not interfere with clinical routine. In lin with this notion, the intervention is chosen by the treating physician in a shared decision making process involving the patient
  Groups: Episodic Migraine

SUMMARY:
This study aims to improve the pathophysiological understanding of migraine in in a longitudinal observational study investigating changes of established neurophysiological and imaging parameters in line with changes of the clinical phenotype.

The study's focus is the investigation of mechanisms that are directly related to the cyclic character of migraine and its core structures. In this context, the primary endpoint is a change in the nociceptive blink reflex, an established brain stem reflex to study the trigemino-spinal system, associated with changes in migraine frequency and severity. In order to reliably detect changes in the trigeminal pain system, investigations are performed in patients before starting a prophylactic therapy and 3 months afterwards. Several secondary endpoints are used to evaluate changes of multimodal sensory and cortical information processing. Cerebral imaging will include examinations of structural and network effects of altered migraine disease activity.

ELIGIBILITY:
Inclusion Criteria (migraineurs):

* episodic migraine according to ICHD (international classification of headache disorders)-3 criteria
* headache documented over at least 3 months through a headache calender
* scheduled for prophylactic therapy of their migraine

Exclusion Criteria (migraineurs):

* history of chronic migraine
* current medication-overuse headache
* neurological or psychiatric diagnosis other than headaches
* chronic intake of central nervous system active drugs (antidepressants, antipsychotics etc.)
* contraindications for magnetic resonance imaging
* contraindications for transcranial magnetic stimulation

Inclusion criteria (controls):

* not more than 3 years younger or older than matched control
* gender similar to matched control
* menstrual cycle equal to matched control (if female)

exclusion criteria (controls):

* more than 1 headache day/month
* history of migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients seen in the local headache clinic are screened for eligibility to participate the study. Clinical routine is not influenced by participation in this observational study, importantly choice of prophylactic treatment solely depends on the physician's and patient's decision based on national guidelines.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
nociceptive blink reflex habituation | baseline and after 3 months
  habituation of the area under of the curve of the R2 blink reflex component on the side primarily affected by migraine headaches

SECONDARY OUTCOMES:
nociceptive blink reflex area | baseline and after 3 months
  area under of the curve of the R2 blink reflex component on the side primarily affected by migraine headaches
somatosensory evoked potentials (SSEP) | baseline and after 3 months
  habituation of the N20 SSEP component following bilateral median nerve stimulation
pattern-reversal visual evoked potentials (VEP) | baseline and after 3 months
  habituation of the P100 VEP component following bilateral optic nerve stimulation
migraine headache frequency | baseline and after 3 months
  days with migraine headaches during the last month
headache impact test (HIT-6) | baseline and after 3 months
  impact of migraine severity on daily routine
migraine disability assessment (MIDAS) | baseline and after 3 months
  impact of migraine frequency on daily routine
Patient-Reported Outcomes Measurement Information System Profile 29 (PROMIS-29) | baseline and after 3 months
  multi domain patient reported quality of life

OTHER OUTCOMES:
transcranial magnetic stimulation (TMS) | baseline and after 3 months
  input-output curves of motor evoked potential following single and double-pulse navigated TMS to the side stimulated during the nociceptive blink reflex examination
electroencephalography (EEG) | baseline and after 3 months
  EEG connectivity following nociceptive and sensory stimulation
structural magnetic resonance imaging (sMRI) | baseline and after 3 months
  volumetry of brain structures involved in central pain processing (e.g. cingulate cortex, insula, thalamus)
functional magnetic resonance imaging (fMRI) | baseline and after 3 months
  resting-state connectivity of networks involved in central pain processing

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Thiele A, Klehr L, Strauss S, Angermaier A, Schminke U, Kronenbuerger M, Naegel S, Fleischmann R. Preventive treatment with CGRP monoclonal antibodies restores brain stem habituation deficits and excitability to painful stimuli in migraine: results from a prospective case-control study. J Headache Pain. 2021 Dec 11;22(1):149. doi: 10.1186/s10194-021-01364-x. PMID 34895133